CLINICAL TRIAL: NCT05299021
Title: The Analgesic Effect of Ultrasound-guided Double-point Versus Single-point Serratus Anterior Plane Block on Modified Radical Mastectomy：A Randomized Controlled Study
Brief Title: Serratus Anterior Plane Block for Modified Radical Mastectomy: Double-point VS Single-point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Director of the department of anaesthesiology, Shanghai cancer center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAPB for MRM 2.0
Record Dates: First submitted 2021-12-06; First posted 2022-03-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-12

CONDITIONS: Mammary Cancer; Serratus Anterior Plane Block; Postoperative Pain
Keywords: Mammary Cancer; Serratus Anterior Plane Block; Postoperative Pain; Axillary Discomfort
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-point SAPB (Experimental): SAPB will be performed simultaneously in both the third and fifth rib levels.
  Interventions: Procedure: Double-point SAPB
- Single-point SAPB (Experimental): SAPB will be performed only in the fifth rib level.
  Interventions: Procedure: Single-point SAPB

INTERVENTIONS:
Procedure: Double-point SAPB — A high-frequency linear probe (6-13 MHz) of the ultrasound machine was used to identify the fifth rib in the midaxillary line. The anatomic landmarks of the block were identified: latissimus dorsi, serratus anterior, and the intercostal muscles in the fourth and fifth intercostal levels. After sterilization and draping, an 20-gauge needle was introduced craniocaudally using an in-plane technique. The needle tip was advanced, targeting the plane between the serratus anterior muscle and the fifth rib. Needle position was confirmed by injection of 1-to-2 mL of saline after negative aspiration. And use the same method targeting the plane between the serratus anterior muscle and the third rib.Under real-time visualization, total 30 mL of 0.375% ropivacaine and 0.5 μ g/kg dexmedetomidine mixture will be injected into the two points with 15 ml separately.
  Arms: Double-point SAPB
Procedure: Single-point SAPB — A high-frequency linear probe (6-13 MHz) of the ultrasound machine was used to identify the fifth rib in the midaxillary line. The anatomic landmarks of the block were identified: latissimus dorsi, serratus anterior, and the intercostal muscles in the fourth and fifth intercostal levels. After sterilization and draping, an 20-gauge needle was introduced craniocaudally using an in-plane technique. The needle tip was advanced, targeting the plane between the serratus anterior muscle and the fifth rib. Needle position was confirmed by injection of 1-to-2 mL of saline after negative aspiration.Under real-time visualization, total 30 mL of 0.375% ropivacaine and 0.5μ g/kg dexmedetomidine mixture will be injected.
  Arms: Single-point SAPB

SUMMARY:
Nowadays, the incidence of breast cancer is the first number of malignant tumors, and the primary treatment method is surgery. As is known to all, less postoperative complications and enhanced recovery are closely related to effective analgesia. However, postoperative patients often experience moderate pain, while associated with axillary discomfort. Serratus Anterior Plane Block (SAPB) relieves postoperative pain, but traditional single point block method has no effect on axillary discomfort. Therefore, it is necessary to try double point blocks to explore their impact on postoperative analgesia and axillary comfort. This RCT will recruit patients proposed to undergo Modified Radical Mastectomy (MRM) and be randomized to single point or double point groups to evaluate their postoperative pain score and axillary comfort in order to provide clinical guidance.

DETAILED DESCRIPTION:
The conventional SAPB, which often performs single point block from the level of the fifth rib, does not completely relieve postoperative pain in patients with axillary lymph node dissection, probably due to insufficient range of local anesthetic diffusion.Anatomical study indicated that with a double point SAPB at the third and fifth rib levels, respectively, the local anesthetic diffusion range can reach the axillary level and may provide better analgesic effects. However, the support of clinical data is lacking.Therefore, the hypothesis of this study is that double point SAPB will provide better postoperative analgesia compared with conventional single point SAPB in patients undergoing modified radical mastectomy.This study will include 60 patients proposed to undergo modified radical mastectomy, allocated to the Double-point or Single-point group in a 1:1 ratio, randomly.The Double-point group will perform a double point SAPB, which is a combined block at the third and fifth rib levels, respectively.The Single-point group will undergo a single point SAPB, traditionally performed at the level of the fifth rib.Observation outcomes included changes in blood pressure and heart rate during dissection of skin and dissection of axillary lymph nodes, postoperative pain scores, axillary comfort, recovery quality, and related complications and postoperative hospital stay.Therefore, the objective is to investigate whether this simple technical modification can better reduce postoperative pain and promote rehabilitation in patients with modified radical mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients are proposed to undergo Modified Radical Mastectomy
* Patients with American Society of Anesthesiologists (ASA) physical status I~III
* aged 18-70 years
* BMI ≤ 35 kg/m2

Exclusion Criteria:

* Patients with a pre-existing neuropathy or sensory deficit affecting the operative region
* Pregnancy
* Chronic pain or opioid dependence (at least 30 mg of oxycodone or equivalent per day)
* Allergy to local anaesthesia or any component of the proposed multimodal analgesia regimen
* Local or systemic contra-indications to peripheral nerve blocks (local infection at the puncture site, coagulopathy, platelets less than 80*10^9/L and prothrombin time more than 15 s)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer patients
Enrollment: 57 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain severity at 24 h | 24 hours after the surgery
  Postoperative pain severity at rest and movement measured using a numerical rating scale(NRS) at 24 h. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side.

SECONDARY OUTCOMES:
Pain severity at discharge from PACU and at 6 and 12 and 48 h postoperatively | Respectively at discharge from PACU and at 6 and 12 and 48 h after the surgery;
  Secondary analgesic outcomes included: pain severity at rest and movement measured using a NRS at discharge from PACU and at 6 and 12 and 48 h postoperatively;
Postoperative opioid consumption | Respectively at 24 and 48 h after the surgery;
  At the end of surgery, patients use postoperative controlled analgesia pump, equip with 0.75 μg / ml sufentanil without background dose, locking time is 10min, and each controlled dose is 2 ml. The cumulative amount of sufentanil used at 24 and 48 hours after surgery will be recorded separately.
Proportion of rescue analgesia | 48 h after the surgery;
  Rescue analgesia was started when NRS ≥ 4, with Flurbiprofen Axetil 50mg i. v. The proportion of patients who required at least one rescue analgesia at 48 hours after surgery will be recorded.

OTHER OUTCOMES:
Postoperative axillary comfort severity | Respectively at discharge from PACU and at 6 and 12 and 24 and 48 h after the surgery.
  Referring to the pain numerical rating scale, make the axillary comfort numerical rating scale. An integer of 0 to 10 is used to indicate different levels of axillary discomfort, and "0" is "no discomfort", and "10" is the "most severe axillary discomfort".Patients are instructed to circle the number that represents the amount of axillary comfort that they are experiencing at the time of the evaluation.
Postoperative quality of recovery | Respectively at 24 and 48 h after the surgery.
  Quality of recovery (QoR) after the surgery will be assessed using a Quality of recovery 15 (QoR-15) scale. This scale is a self-rated patient-centered system for the assessment of the quality of early postoperative recovery, including five dimensions: emotional state, physical comfort, psychological support, physiological independence and pain, with 15 items and scores ranging from 0 to 150, and higher scores indicate a better quality of postoperative recovery.
Changes in mean arterial pressure（MAP） and heart rate during skin peeling and axillary node dissection | Before and after 3 min of incision, before and after 3 min of axillary lymph nodes,respectively.
  Perfect analgesia can reduce the effect of surgical stimulation on heart rate and MAP. Surgical stimulation increases at the onset of peeling or the dissection of the axillary lymph nodes, when the magnitude of changes in MAP and heart rate can indirectly reflect the degree of analgesia.MAP and heart rate will be therefore recorded before and after 3 min of incision, before and after 3 min of axillary lymph nodes respectively.
Proportion of postoperative nausea and vomiting | up to 48 hours postoperatively.
  Proportion of patients experiencing postoperative nausea and vomiting at least once at 48 h postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Ling D, Xu Q, Sun P, Wei S, Gao L, Lou F, Zhang J. Ultrasound-Guided Double-Point Versus Single-Point Serratus Anterior Plane Block for Modified Radical Mastectomy: A Randomized Controlled Trial. Clin J Pain. 2025 Jan 1;41(1):e1256. doi: 10.1097/AJP.0000000000001256. PMID 39475834